CLINICAL TRIAL: NCT07297264
Title: Effect of Betamethasone Injection Into the Pterygomandibular Space on Postoperative Sequelae of Impacted Lower Third Molar Surgery: A Randomized, Double-blind, Placebo-controlled Clinical Trial With a Split-mouth Design
Brief Title: Betamethasone and Complications of Lower Third Molar Surgery
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: There was a change in the protocol of the study
Sponsor: Shehab Ahmed Hamad (Other)
Responsible Party: Sponsor-Investigator, Shehab Ahmed Hamad, Assisstan professor, Kurdistan Higher Council of Medical Specialties
Organization: Kurdistan Higher Council of Medical Specialties (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: Betamethasone in MTM
Record Dates: First submitted 2023-04-19; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Morbidity; Third Molars Extraction; Steroid Injection
MeSH Terms: interventions — Betamethasone; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- betamethasone treated side (Experimental): Betamethasone was administered into the pterygomandibular space immediately before surgery
  Interventions: Drug: Betamethasone
- Control side (Placebo Comparator): normal saline was administered into the pterygomandibular space immediately before surgery
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Betamethasone — The study group (group I) received 1 ml (6 mg) of betamethasone (CKOÇAK FARMA, Turkey) injection to the pterygomandibular space. Each ml contains 3.0 mg betamethasone acetate and 3.0 mg betamethasone sodium phosphate
  Other Names: Betamethasone injection ino the pterygomandibular space
  Arms: betamethasone treated side
Drug: normal saline — normal saline
  Arms: Control side

SUMMARY:
Pain, swelling, and trismus are common sequalae of surgical removal of impacted third molars. The aim of this study is to evaluate effect of local administration of betamethasone, into the pterygomandibular space, on these sequalae

DETAILED DESCRIPTION:
A prospective, single center, double-blind, randomized controlled design study was conducted between January 2022 and February 2023, in the department of oral and maxillofacial surgery, Rizgary teaching hospital, Erbil, Iraq. The participants were patients presented for the surgical removal of bilateral symmetrical impacted lower third molars. To achieve 95% power, a sample size of 40 patients with bilateral impacted third molars was required.

The study was approved by the Ethical Committee of the institutional board and was conducted in accordance with the guidelines of the World Medical Association Declaration of Helsinki (1964) and its seventh amendment (2013) and to the Consolidated Standards of Reporting Trials (CONSORT) (Figurec1). The objectives of the study, as well as the risks and benefits were explained to the patients and those who agreed to participate have signed a consent form.

The inclusion criteria of the study were: individuals of both genders aging between 18 and 35 years, classified as ASA I according to the American Society of Anesthesiologists, and who have symmetrical bilateral impacted mandibular third molar detected by a panoramic radiograph. Impacted teeth categorized as mesiaoangular (Winter classification) and class II position B (Pell and Gregory classification) were included. The patients had no infection, pain, trismus, and swelling at the time of surgery.

Patients who are smokers, with pericoronitis, active infection, systemic disorders, on long term steroids, pregnant and lactating women were excluded. Patients were also precluded if they had taken analgesics 24 hours before- and antibiotics one week before the surgery, and if the surgical procedure exceeded 30 minutes or if more than three cartridges of local anaesthesia were used during the procedure.

By implementing the split mouth model, each participant underwent two surgical procedures, with an interval of at least 4 weeks between them. Prior to the first procedure, randomization of the first side to be operated (right or left) was performed using the "heads or tails" technique using a coin, where the head represented the right side and tails the left side.

The study group (group I) received 1 ml (6 mg) of betamethasone (CKOÇAK FARMA, Turkey) injection to the pterygomandibular space. Each ml contains 3.0 mg betamethasone acetate and 3.0 mg betamethasone sodium phosphate. The control group (group II) received a corresponding volume of normal saline injected into the pterygomandibular space. To ensure blinding of the study, the solution was injected by a third person, who is not directly involved in the surgery nor in the postoperative visits.

Impacted mandibular third molar surgery was performed under local anesthesia, using 2% lidocaine hydrochloride with 1:80,000 concentration of adrenaline. Inferior alveolar nerve, lingual and buccal nerve block technique were performed. After profound anesthesia was achieved, the betamethasone, or the sham solution, was injected into the pterygomandibular space using 3 ml disposable plastic syringe and gauge 25 hypodermic needle. A standard Ward's incision was designed and the mucoperiosteal fap was reflected to expose the surgical site. A lingual flap was reflected, only when deemed to be necessary. Bone guttering was made using round No.8 and straight fissure carbide bur (no. 703) bur, under copious saline irrigation. The tooth was sectioned or removed as whole. It was then luxated and delivered using elevators and forceps. The socket was thoroughly irrigated with normal saline solution done, after the rough bone margins were trimmed and finally the wound was closed with 3-0 Vicryl suture. The duration of surgery was measured from the time of incision to placement of the last suture.

The patient was given the usual postoperative instructions, including ice pack application to the operated side for 20 minutes, with 20-minute intervals between applications, for the first day. The patient was advised to consume cold liquid diet in the first day, and soft diet for the next 5 days. In addition, twice daily mouth wash with chlorhexidine 0.12% for 5 days, starting the day after surgery. Patients were given three days course of broad-spectrum antibiotic (amoxicillin 500 mg every eight hours or clindamycin 300 mg every eight hours if a penicillin allergy existed) and paracetamol 1g as a rescue analgesic.

The Facial swelling and the degree of trismus was recorded by the same operator, preoperatively and on the first, third, and seventh postoperative days. The pain was recorded by the patient, at 8:00 am, using visual analogue scale (VAS) at 1-5 postoperative days. . The patients rated pain on a 10-cm VAS, from no pain (0) to the most severe pain (10). Number of analgesic tablets consumed by the patients ,during the first five postoperative days, was also calculated. Flexible tape was used for measuring the following facial distances: gonion-lip commissure, gonion-external canthus of the eye, tragus-lip commissure, tragus-soft tissue pogonion. The sum of the preoperative measurements was considered as a baseline for the side of the face being assessed. Subtracting the preoperative measurement from the postoperative one indicated the amount of facial swelling. The degree of trismus was assessed by measuring the distance between the incisal edges of the upper and lower central incisors, on maximum mouth opening, using a digital vernier Statistical analyses was performed using the statistical package SPSS software 25.0. Comparisons between the groups was carried out using an independent t test. The significance level was set at P < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* no infection
* no pain
* no limitation of mouth opening
* symmetrical bilateral impacted third molars (Mesioangular, CLASS II, Position B

Exclusion Criteria:

* Infection
* systemic disease
* smokers
* operation time exceeding 30 minutes

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-01-03 (Actual); Primary Completion 2023-02-21 (Actual); Study Completion 2023-03-26 (Actual)

PRIMARY OUTCOMES:
Postoperative pain was assessed by patient self-report using a visual analogue scale (VAS; 0-10), where 0 indicated no pain and 10 indicated the worst imaginable pain. | Pain scores were recorded immediately after surgery and daily for the first five days
  postoperative pain assessed by the patient on VAS pain score

SECONDARY OUTCOMES:
trismus | Trismus was measured on the first, third, and seventh postoperative days
  degree of maximum mouth opening measured between the maxillary and mandibular central incisors using a digital vernier
Facial swelling | Facial swelling was measured on the first, third, and seventh postoperative days
  Flexible tape was used for measuring the following facial distances: gonion-lip commissure, gonion-external canthus of the eye, tragus-lip commissure, tragus-soft tissue pogonion. The sum of the preoperative measurements was considered as a baseline for the side of the face being assessed. Subtracting the preoperative measurement from the postoperative one indicated the amount of facial swelling.

CONTACTS AND LOCATIONS:
Overall Officials: Shehab Hamad, FFDRCSI, Principal Investigator — Kurdistan Higher Council of Medical Specialties
Locations (1):
- Shehab Ahmed Hamad, Erbil, Iraq